CLINICAL TRIAL: NCT04483375
Title: A Randomized, Double-blinded, Placebo-controlled, Single Ascending Dose, Phase I Study to Evaluate the Tolerability, Safety, Pharmacokinetics of SCTA01 in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of SCTA01, an Anti-SARS-CoV-2 Monoclonal Antibody, in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCTA01-X101
Record Dates: First submitted 2020-07-17; First posted 2020-07-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus Disease 2019(COVID-19)
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — upanovimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-SARS-CoV-2 monoclonal antibody(SCTA01) (Experimental): SCTA01: single dose on Day0
  Interventions: Biological: SCTA01
- Placebo (Placebo Comparator): Placebo: single dose on Day0
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SCTA01 — recombinant humanized anti-SARS-CoV-2 monoclonal antibody
  Arms: anti-SARS-CoV-2 monoclonal antibody(SCTA01)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety, pharmacokinetics of SCTA01(anti-SARS-CoV-2 monoclonal antibody) in Healthy Chinese Subjects.

DETAILED DESCRIPTION:
This is a Phase 1, First-in-Human, Randomized, Double-blinded, Placebo-Controlled, Single Ascending Dose Study of SCTA01(Anti-SARS-CoV-2 monoclonal antibody) in Healthy Chinese Subjects.

Dose escalation will be guided by a safety review of clinical signs and symptoms, adverse events (AEs), and laboratory results of the prior dose cohort.

An Interim analysis will be performed after Day 28 post-dose for the last dose cohort for review.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Males or females. Aged ≥ 18 years old
* Body mass index (BMI) between 18.0 and 26.0 kg/m2
* Normal or abnormal but non-clinical significant physical examination, vital signs, 12-ECG and chest CT, etc
* No plan of pregnancy and being willing to use effective contraceptive measures (including partner) from informed consent to 6 months after administration of SCTA01/placebo (abstinence，sterilization operation，contraceptive barrier，acyeterion , etc.)

Exclusion Criteria:

* Having a history of severe allergy, such as severe allergic reactions, urticaria, angioedema;
* Having one of the following evidence on SARS-CoV-2 infection(previous tests were accepted)：

  * SARS-CoV-2 positive: reverse transcription-polymerase chain reaction (RT-PCR) and/or next generation sequencing (NGS)
  * Previous viral gene sequencing showed high homology with the known SARS-CoV-2
  * Positive specific antibody IgM or IgG against serum SARS-CoV-2
* Having a history of severe allergies, such as severe allergic reactions, urticaria, angioedema;
* Having active infection or fever before to enrollment(≥ 37.3℃)
* Having primary disease in main organs, such as heart, lung, kidney, liver, nervous system, gastrointestinal system dysfunction, history of thrombocytopenia or abnormal bleeding
* Suffering from autoimmune diseases or a history of autoimmune diseases (such as systemic lupus erythematosus, thyroid Inflammation, vasculitis, etc.)
* Within 7 days prior to the first dose of SCTA01/placebo, subject has received any prescription drugs, non-prescription drugs, Chinese herbal medicines and health products
* Within 3 months prior to the first dose of SCTA01/placebo, subjects who participated in other clinical study, or remaining in the elimination period of the drug (within 5 half-lives) before treatment
* Within 30 days prior to the first dose of SCTA01/placebo, subjects who have received vaccine
* Within 3 months prior to the first dose of SCTA01/placebo, subjects who have received blood product treatment or blood donation and hemorrhage ≥400mL, or subjects who has a blood donation plan within 3 months after treatment
* Within 6 months prior to the first dose of SCTA01/placebo, subjects who have received major surgery, or has surgery plan during clinical trail
* Pregnant or lactating women or positive β-HCG, has plan of pregnancy from informed consent signed to 6 months after administration of SCTA01/placebo
* Positive of anti-HIV, TP-Ab, anti-HCV, anti-HBV
* Having a history of epilepsy
* Having a history of malignancies
* Within 3 months prior to screening, sujects who have drunk more than 14 standard units (1 standard unit contains 14g alcohol, such as 360mL beer, 45mL spirits with 40% alcohol or 150mL wine), or positive of alcohol breath test
* Within 3 months prior to screening, subjects who smoked more than 5 cigarettes per day, do not accept smoking cessation during the study
* Having a history of drug addiction and drug abuse; or who have a positive urine test result for drug abuse; or cannot guarantee that they will not abuse drugs during the study
* Subjects who are not able to follow the plan to complete the study
* Subjects who are not considered suitable for the study by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 7 days
  DLT will be assessed by DAIDS v2.1. The measurements include clinical symptoms and abnormal vital signs, abnormal laboratory tests (complete blood cell count, serum chemistry, routine urinalysis, coagulation function, etc.) and 12-lead ECGs
Maximal Tolerable Dose(MTD) | 12 weeks
  MTD will be assessed by DAIDS v2.1. The measurements include clinical symptoms and abnormal vital signs, abnormal laboratory tests (complete blood cell count, serum chemistry, routine urinalysis, coagulation function, etc.) and 12-lead ECGs.

SECONDARY OUTCOMES:
AUC0-t | 12 weeks
  Area under the curve from the time of dosing to the last measurable concentration time t (AUC0-t)
AUC0-∞ | 12 weeks
  Area Under the Concentration Time Curve (AUC) From Time Zero to Infinity (AUC 0-∞)
t1/2 | 12 weeks
  Elimination Phase Half-life(t1/2)
Tmax | 12 weeks
  Time to the Maximum Concentration(Tmax)
Anti-drug antibody(ADA) | 12 weeks
  Positive rate of anti-SCT A01 antibody
Adverse events | 12 weeks
  Adverse events as assessed by DAIDS v2.1, including clinical symptoms and abnormal vital signs, abnormal laboratory tests (complete blood cell count, serum chemistry, routine urinalysis, coagulation function, etc.) and 12-lead ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Xinghe Wang, MD,PhD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing SHIJITAN Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Li Y, Qi L, Bai H, Sun C, Xu S, Wang Y, Han C, Li Y, Liu L, Cheng X, Liu J, Lei C, Tong Y, Sun M, Yan L, Chen W, Liu X, Liu Q, Xie L, Wang X. Safety, Tolerability, Pharmacokinetics, and Immunogenicity of a Monoclonal Antibody (SCTA01) Targeting SARS-CoV-2 in Healthy Adults: a Randomized, Double-Blind, Placebo-Controlled, Phase I Study. Antimicrob Agents Chemother. 2021 Oct 18;65(11):e0106321. doi: 10.1128/AAC.01063-21. Epub 2021 Sep 7. PMID 34491805
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343